CLINICAL TRIAL: NCT00186719
Title: How Smoking Causes COPD: Examination of Immune System Changes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Gerard Cox, St. Joseph's Healthcare Hamilton
Other Study IDs: 02-2182
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Smoking Related Disease; Immune System Changes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A breathing condition known as "chronic obstructive pulmonary disease" (COPD) caused by cigarette smoking is a major health problem. The way by which smoking leads to lung disease is uncertain. Recent research done in animals provides a description of specific changes (that is a reduction) in these immune cell types as a result of cigarette smoke exposure. The study you have been asked to participate in is a pilot study to see if similar changes occur in humans who smoke. The purpose of this study is to evaluate this new method of testing blood in 3 groups of 10 people: normal non-smoking subjects, subjects who smoke with no history of lung disease and subjects who smoke and have smoking related COPD.

DETAILED DESCRIPTION:
The mechanism by which smoking leads to damage to lung tissue in susceptible hosts, is uncertain. Recently there has been description of specific changes (that is reduction) in the number and activity of certain key immune cell types - dendritic cells- as a result of cigarette smoke exposure. This work was done in animal models and we would like to develop methods that will allow us to examine if similar changes occur in humans who smoke. Reduced number and activity of dendritic cells would be expected to lead to increased incidence of infection - a common problem in patients with COPD.

Since dendritic cells come to the lung from the bloodstream, and one can detect them in the circulation, we will look at the dendritic cells that are present in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* Healthy Subjects - Non smokers
* FEV1/FVC > 70% predicted
* Current Smokers - > 10 pack year smoking history
* FEV1/FVC > 70% predicted
* Current Smokers with COPD - > 10 pack year smoking history
* FEV1/FVC < 70% predicted
* Able to give informed consent

Exclusion Criteria:

* Healthy Subjects - Reside with smokers
* History of lung disease
* Current Smokers - History of lung disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: smokers and non-smokers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Study Completion 2012-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cox, MB FRCPC FRCPI, Principal Investigator — McMaster University
Locations (1):
- St Joseph's Healthcare, Hamilton, Ontario, Canada